CLINICAL TRIAL: NCT01319097
Title: Clinical Study of Evaluate the Effect of Sorbion Sachet S Wound Dressing on Soft Tissue Edema and Wound Bioburden in Moderately to Highly Exuding Pressure Ulcers
Brief Title: Study to Evaluate the Effect of Sorbion Sachet S Wound Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Regional Wound Care Center (Other)
Collaborators: Sorbion Aktiengesellschaft, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56-RW-017
Record Dates: First submitted 2011-03-09; First posted 2011-03-21 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Pressure Ulcers
Keywords: Reduction on local soft tissue edema
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorbion Sachet S (Other): Subject will evaluate Sorbion Sachet S dressing for 4 weeks.
  Interventions: Other: Sorbion Sachet S

INTERVENTIONS:
Other: Sorbion Sachet S — Dressing is indicated for moderately to heavily exuding wounds.

SUMMARY:
This is a clinical study to evaluate the effects of sorbion sachet s wound dressing on soft tissue edema and wound bioburden in moderately to highly exuding pressure ulcers.

DETAILED DESCRIPTION:
This study is aimed at the participation of subject with moderately to highly exuding pressure ulcers. Each Subject is expected to participate for a period of 4 weeks or until reepithelization, which occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Subject > 18 years.
* Subject is attending SW Wound Care Center
* Subject has a wound not smaller than 1cm2
* Subject has a wound not larger than 14cm X 23cm
* Subject has a moderately to highly exudative pressure ulcer that would be indicated for treatment with sorbion sachet S
* Subject or subject's legally authorized representative is informed about the trial, understands the nature of the study and provides written informed consent prior to study enrollment.
* Subject is willing and able to comply with all specified care and visit requirements.

Exclusion Criteria:

* Subject has a lesion that does not meet the inclusion criteria.
* Subject has a pressure ulcer that contains areas of undermined tissue.
* Subject refuses to participate in the study.
* Subject is participating in another clinical study.
* Subject already participates in this study with one wound (only one wound per subject is allowed)
* Subject has known sensitivity to the trial product or any of its compounds.
* Subject is expected to be non-compliant.
* Subject uses therapy known to be immunocompromising such as systemic anti cancer drugs and/or systemic corticosteroids.
* Subject suffers from systemic infectious disease(s) known to negatively influence wound healing, such as AIDS.
* Subject's lesion is a primary skin cancer.
* Subject's lesion is the manifestation of a metastasis.
* Subject is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate the effect of sachet S reduction on local soft tissue edema (excessive interstitial fluid to a maximum 3cm depth) in pressure ulcers. | 1 year
  To investigate the effect of sachet S reduction on local soft tissue edema in pressure ulcers and the degree to which sachet S influences the wound surface bioburden qualitatively and quantitatively.

SECONDARY OUTCOMES:
The secondary objectives are to further investigate whether sorbion sachet s | 1 year
  Generates changes in subjective parameters Generates changes in wound size Leads to clinician satisfaction and patient compliance with sachet s

CONTACTS AND LOCATIONS:
Overall Officials: Randall D Wolcott, M.D., Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States